CLINICAL TRIAL: NCT05706649
Title: Effect of Plant-based Diet on Postprandial Sleepiness
Brief Title: A Study of Plant-based Diet on Postprandial Sleepiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph Y. Cheung, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22-011794
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Drowsiness
Keywords: Postprandial Sleepiness
MeSH Terms: conditions — Sleepiness | interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant-based diet (Experimental): Subjects will receive a handbook on plant-based diet including recipe recommendations. They will follow a strict plant-based diet for 21 day.
  Interventions: Behavioral: Plant-based diet

INTERVENTIONS:
Behavioral: Plant-based diet — 21 day diet that excludes any form of meat and other animal products, including dairy products.

SUMMARY:
This research aims to develop a better understanding and clinical knowledge of the effects of a plant-based diet on postprandial sleepiness.

ELIGIBILITY:
Inclusion Criteria

* Sleepiness after eating lunch.
* ESS score ≥3 for answering the question about these two situations: 'sitting quietly after lunch without alcohol' and 'lying down to rest in the afternoon when circumstances permit'.

Exclusion Criteria

* Diabetes.
* Pregnancy or lactation.
* Current use of a vegan/plant-based diet
* BMI ≤ 22.
* Iron deficiency.
* Vitamin B12 deficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Change in postprandial sleepiness | Baseline, 21 days
  Measured by Epworth Sleepiness Questionnaire before and after a plant-based diet. The Epworth sleepiness scale (ESS) is an 8 item questionnaire that measures daytime sleepiness in participants. Possible scores range from 0-24, with higher scores indicating a higher average sleep propensity in daily life, and a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheung, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials